CLINICAL TRIAL: NCT00003941
Title: A Randomized Phase III Study of Sequential High-Dose Cisplatinum/Etoposide/Ifosfamide Plus Stem Cell Support Versus BEP in Patients With Poor Prognosis Germ Cell Cancer
Brief Title: Combination Chemotherapy With or Without Peripheral Stem Cell Transplant in Treating Men With Previously Untreated Germ Cell Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Allocation: Randomized | Purpose: Treatment
Other Study IDs: EORTC-30974; EORTC-30974
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2012-09-24 (Estimated); Status verified 2012-09

CONDITIONS: Mediastinal Cancer; Metastatic Cancer; Testicular Germ Cell Tumor
Keywords: stage III malignant testicular germ cell tumor; mediastinal cancer; testicular embryonal carcinoma; testicular choriocarcinoma; testicular teratoma; testicular yolk sac tumor; testicular embryonal carcinoma and teratoma; testicular embryonal carcinoma and teratoma with seminoma; testicular embryonal carcinoma and yolk sac tumor; testicular embryonal carcinoma and yolk sac tumor with seminoma; testicular embryonal carcinoma and seminoma; testicular yolk sac tumor and teratoma; testicular yolk sac tumor and teratoma with seminoma; testicular choriocarcinoma and yolk sac tumor; testicular choriocarcinoma and embryonal carcinoma; testicular choriocarcinoma and teratoma; testicular choriocarcinoma and seminoma; tumors metastatic to brain; liver metastases; bone metastases
MeSH Terms: conditions — Mediastinal Neoplasms; Neoplasm Metastasis; Testicular Germ Cell Tumor; Testicular Neoplasms; Teratoma, Testicular; Endodermal Sinus Tumor; Teratoma; Seminoma; Carcinoma, Embryonal; Brain Neoplasms | interventions — Bleomycin; Filgrastim; Cisplatin; Etoposide; Ifosfamide; Peripheral Blood Stem Cell Transplantation

INTERVENTIONS:
Biological: bleomycin sulfate
Biological: filgrastim
Drug: cisplatin
Drug: etoposide
Drug: ifosfamide
Procedure: bone marrow ablation with stem cell support
Procedure: peripheral blood stem cell transplantation

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Combining more than one drug may kill more cancer cells. Peripheral stem cell transplant may allow the doctor to give higher doses of chemotherapy and kill more cancer cells. It is not yet known whether chemotherapy and peripheral stem cell transplant is more effective than chemotherapy alone.

PURPOSE: This randomized phase III trial is studying how well combination chemotherapy works when given with peripheral stem cell transplant and how it compares with combination chemotherapy alone in treating men with previously untreated germ cell cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the efficacy of standard cisplatin, etoposide, and ifosfamide (VIP) followed by sequential high-dose VIP and stem cell rescue versus bleomycin, etoposide, and cisplatin (BEP) in men with previously untreated poor-prognosis germ cell cancer.
* Compare the acute and late toxicities of these treatment regimens in this patient population.
* Compare these regimens in terms of failure-free survival, response rate, and overall survival in these patients.
* Evaluate the quality of life in these patients.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to center, primary mediastinal germ cell tumor (yes vs no), and nonpulmonary visceral metastases (liver vs bone vs brain). Patients are randomized to one of two treatment arms.

* Arm I: Patients receive etoposide IV over 1 hour followed by cisplatin IV over 1 hour on days 1-5 and bleomycin IV over 30 minutes on days 2, 8, and 15. Treatment repeats every 3 weeks for 4 courses.
* Arm II: Patients receive 1 course of standard dose chemotherapy consisting of etoposide IV over 1 hour followed by cisplatin IV over 1 hour and ifosfamide IV over 1 hour on days 1-5. Peripheral blood stem cells (PBSC) are harvested around day 12-15. Patients also receive daily filgrastim (G-CSF) subcutaneously beginning on day 6 and continuing until PBSC collection is complete.

After day 21, patients receive high-dose chemotherapy consisting of etoposide IV over 1 hour followed by cisplatin IV over 1 hour, and ifosfamide IV over 1 hour on days -6 through -2. PBSCs are infused on day 0. Patients receive daily G-CSF subcutaneously beginning on day 1 and continuing through day 19 or until blood counts have recovered. Treatment repeats every 3 weeks for 3 courses in the absence of disease progression or unacceptable toxicity.

Quality of life is assessed before chemotherapy, at 6 months, and at 2 years after treatment.

Patients are followed monthly for 1 year, every 2 months for 1 year, every 3 months for 1 year, every 6 months for 1 year, and annually thereafter.

PROJECTED ACCRUAL: A total of 222 patients (111 per treatment arm) will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven germ cell cancer

  * Nonseminoma OR
  * Combined seminoma and nonseminoma
* Poor prognosis (nonseminoma):

  * Testis/retroperitoneal primary AND
  * One of the following poor tumor markers

    * AFP greater than 10,000 iu/L
    * HCG greater than 50,000 iu/L
    * LDH greater than 10 times upper limit of normal OR
  * Nonpulmonary visceral metastases (i.e., liver, bone, or brain) OR
  * Mediastinal primary

PATIENT CHARACTERISTICS:

Age:

* 16 to 50

Sex:

* Male

Performance status:

* WHO 0-3

Life expectancy:

* Not specified

Hematopoietic:

* WBC at least 3,000/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin no greater than 1.25 times upper limit of normal (ULN)
* AST no greater than 2 times ULN

Renal:

* Creatinine clearance at least 60 mL/min (unless due to obstructive uropathy correctable by nephrostomy)

Other:

* No other malignancy except basal cell skin cancer
* No neuropathy
* No other serious illness or medical condition
* No psychological, familial, sociological, or geographical condition that would prevent compliance

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No prior chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* Concurrent radiotherapy for brain metastases allowed

Surgery:

* Concurrent surgery for brain metastases allowed

Ages: 16 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 222 (Estimated)
Dates: Start 1999-04; Primary Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Failure-free survival as measured by Logrank at 1 year

SECONDARY OUTCOMES:
Complete response as measured by negative tumor markers and no residual masses or viable cancer cells at the end of CT scan or debulking surgery
Overall survival as measured by Logrank at 2 years
Quality of life as measured by Quality of Life Questionnaire-Core 30 (QLQ-C30) v3.0 at baseline, at month 6, and at year 2
Toxicity as measured by NCI-CTC v2.0 after each course, every 6 months up to year 5, and yearly

CONTACTS AND LOCATIONS:
Overall Officials: Gedske Daugaard, MD, DMSc, Study Chair — Rigshospitalet, Denmark
Locations (37):
- Ludwig Boltzmann Institute for Applied Cancer Research at Kaiser Franz Josef Hospital, Vienna (Wien), Austria
- Belgium (3):
  - Institut Jules Bordet, Brussels (Bruxelles)
  - Universitair Ziekenhuis Antwerpen, Edegem
  - U.Z. Gasthuisberg, Leuven
- Denmark (2):
  - Aarhus University Hospital - Aarhus Sygehus - Norrebrogade, Aarhus
  - Rigshospitalet - Copenhagen University Hospital, Copenhagen
- Germany (14):
  - Universitaetsklinikum Bonn, Bonn
  - Staedtisches Klinikum Dessau, Dessau
  - St. Johannes Hospital - Medical Klinik II, Duisburg
  - Universitaetsklinikum Essen, Essen
  - Staedtische Kliniken Frankfurt am Main - Hoechst, Frankfurt
  - Klinik Fuer Innere Medizin, Hematology/Oncology, Ernst Moritz Armdt Universitaet, Greifswald
  - Universitaetsklinikum Halle, Halle
  - Universitaetsklinikum Hamburg-Eppendorf, Hamburg
  - Universitaetsklinikum des Saarlandes, Homburg
  - Knappschaft Krankenhaus, Langendreer
  - Johannes Gutenberg University, Mainz
  - Klinikum Rechts Der Isar - Technische Universitaet Muenchen, Munich (Muenchen)
  - Klinikum Nuernberg - Klinikum Nord, Nuremberg
  - Klinikum der Universitaet Regensburg, Regensburg
- Ospedale di Circolo e Fondazione Macchi, Varese, Italy
- Netherlands (4):
  - Leiden University Medical Center, Leiden
  - Academisch Ziekenhuis Maastricht, Maastricht
  - Universitair Medisch Centrum St. Radboud - Nijmegen, Nijmegen
  - University Medical Center Rotterdam at Erasmus Medical Center, Rotterdam
- Norwegian Radium Hospital, Oslo, Norway
- Maria Sklodowska-Curie Memorial Cancer Center and Institute of Oncology, Warsaw, Poland
- National Cancer Institute - Bratislava, Bratislava, Slovakia
- Spain (6):
  - Hospital de la Santa Cruz i Sant Pau, Barcelona
  - Institut Catala D'Oncologia, Barcelona
  - Hospital Donostia, Donostia / San Sebastian
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Hospital Universitario LA FE, Valencia
  - Hospital Clinico Universitario Lozano Blesa, Zaragoza
- Inselspital Bern, Bern, Switzerland
- United Kingdom (2):
  - Leeds Cancer Centre at St. James's University Hospital, Leeds, England
  - Velindre Cancer Center at Velindre Hospital, Cardiff, Wales

REFERENCES:
- [Result] Daugaard G, Skoneczna I, Aass N, De Wit R, De Santis M, Dumez H, Marreaud S, Collette L, Lluch JRG, Bokemeyer C, Schmoll HJ. A randomized phase III study comparing standard dose BEP with sequential high-dose cisplatin, etoposide, and ifosfamide (VIP) plus stem-cell support in males with poor-prognosis germ-cell cancer. An intergroup study of EORTC, GTCSG, and Grupo Germinal (EORTC 30974). Ann Oncol. 2011 May;22(5):1054-1061. doi: 10.1093/annonc/mdq575. Epub 2010 Nov 8. PMID 21059637